CLINICAL TRIAL: NCT02177526
Title: Detection of Malignant Calcifications in High Grade Prostate Cancer With Comedo-type Necrosis Using Thin Section Computed Tomography and Susceptibility Weighted Magnetic Resonance Imaging
Brief Title: Imaging of High Grade Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: trial logistics
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Malignant Prostate 100
Record Dates: First submitted 2014-06-18; First posted 2014-06-27 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Prostatic Carcinoma
Keywords: CT; MRI
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diagnostic Imaging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imaging - CT and MRI examinations (Other): Abdominal and pelvic CT and pelvic MRI imaging will be performed in 30 patients.
  Interventions: Device: Imaging

INTERVENTIONS:
Device: Imaging — 15 patients with malignant comedo-type necrosis and calcifications detected with histo-pathology from guided biopsies will be enrolled after obtaining informed consent. 15 patients with biopsy proven Gleason pattern 5 tumor and without comedo-type necrosis associated calcification will serve as a comparison group after providing informed consent for a total of 30 patients.
  Other Names: CT; MRI

SUMMARY:
Management of prostatic carcinoma varies according to stage of disease. Trans-rectal ultrasound guided biopsy is known to underestimate the degree of tumor due to undersampling and random non-targeted technique. Methods to improve pre-operative tumor localization and grading, including multi-parametric (MP) magnetic resonance imaging (MRI) is an active area of research but requires further validation.

High grade tumors can undergo comedo-type necrosis with malignant calcifications which only occurs in Gleason pattern 5 tumors and which we hypothesize can be reliably detected using computed tomography (CT) and/or MRI.

Detection of malignant calcification within tumor foci will improve the accuracy of localization and grading in prostatic carcinoma.

DETAILED DESCRIPTION:
High grade (Gleason pattern 5) tumors can undergo comedo-type necrosis producing malignant calcifications which we hypothesize can be reliably detected using computed tomography (CT) and/or MRI. Detection of malignant calcifications in areas of Gleason pattern 5 tumor will improve the accuracy of pre-operative localization and grading in prostatic carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant comedo-type necrosis and calcifications detected with histo-pathology from guided biopsies
* Patients with biopsy proven Gleason pattern 5 tumor and without comedo-type necrosis associated calcification

Exclusion Criteria:

* Patients who do not have malignant comedo-type necrosis and calcifications detected with histo-pathology from guided biopsies

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
The number of prostate patients with comedo-type necrosis. | up to 4 weeks
  Two radiologists will review the MRI and CT examinations separated by a 4 week interval to decrease recall bias. Further, readers will review the 3 additional gradient echo pulse sequences independently at 3 different MRI reading sessions, also separated by 4 weeks, in order to compare the accuracy from each pulse sequence and to reduce recall bias.

SECONDARY OUTCOMES:
The number of other features measured on MRI. | up to 4 weeks
  Two radiologists will review the MRI and CT examinations separated by a 4 week interval to compare other MRI features and clinical factors between Gleason pattern 5 tumors with and without malignant calcification.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Schieda, MD, Principal Investigator — OHRI
Locations (1):
- Ottawa Hospital (Civic Campus), Ottawa, Ontario, Canada